CLINICAL TRIAL: NCT03043807
Title: A Phase II Study of Definitive Therapy for Newly Diagnosed Men With Oligometastatic Prostate Cancer After Prostatectomy
Brief Title: A Study of Definitive Therapy to Treat Prostate Cancer After Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J16151; IRB00120414 (Other: JHU IRB)
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; androgen deprivation; chemotherapy; radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Docetaxel; bicalutamide; Radiation; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- chemohormonal and definitive therapy after prostatectomy (Experimental): (1st) Systemic chemo-hormonal therapy with up to 6-months (~24 weeks) of adjuvant androgen deprivation (Leuprolide Acetate) and up to 6 cycles of chemotherapy (Docetaxel), (2nd) definitive local tumor control with adjuvant radiation therapy, and (3rd) consolidative stereotactic radiation to oligometastatic lesions. The men will receive a total of 2 years of androgen deprivation. Androgen blockade (Bicalutamide) will be the same throughout the course of treatment.
  Interventions: Drug: Leuprolide Acetate; Drug: Docetaxel; Drug: Bicalutamide; Radiation: Radiation; Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Leuprolide Acetate — 22.5mg by intramuscular (IM) injection every 3 months
  Other Names: Lupron Deport
Drug: Docetaxel — 75 mg/m2 IV will be given on day 1 every 3 weeks, up to 6 cycles. Dose may decreased in the following intervals: 65 mg/M2, 55 mg/M2, 35 mg/M2.
  Other Names: Texotere
Drug: Bicalutamide — bicalutamide (Casodex) 50mg by mouth daily
  Other Names: Casodex
Radiation: Radiation — Radiation will be delivered in 1 to 5 fractions, and the dose and fractionation schedule will depend on the size and location of the lesion and the surrounding normal tissue constraints in accordance with AAPM Task Group 101 recommendations. Typical doses include 16 - 24 Gy in 1 fraction, 48 - 50 Gy in 4 fractions, and 50 - 60 Gy in 5 fractions.
Drug: Abiraterone Acetate — Abiraterone acetate 1000 mg / day may be given at the investigator's discretion.
  Other Names: Zytiga

SUMMARY:
To assess the safety of treating men with oligometastatic prostate cancer with the following therapy: (1st) Systemic chemo-hormonal therapy with up to 6-months (~24 weeks) of adjuvant androgen deprivation and up to 6 cycles of chemotherapy, (2nd) definitive local tumor control with adjuvant radiation therapy, and (3rd) consolidative stereotactic radiation to oligometastatic lesions. The men will receive a total of 2 years of androgen deprivation. Androgen blockade will be the same throughout the course of treatment.

DETAILED DESCRIPTION:
Adjuvant treatment (month 1 through ~6): All patients will be treated with up to 6 months of androgen deprivation, plus up to 6 cycles of docetaxel chemotherapy. Following docetaxel therapy, patients with a Prostate-specific antigen response of at least a 50% decrease from baseline, will proceed to maximum consolidative therapy.

Radiation (month 7 though ~11): After completion of adjuvant chemotherapy, the men will be treated with definitive local therapy with adjuvant radiation therapy (RT). After definitive local therapy, patients will be treated with consolidative stereotactic body radiation therapy (SBRT) to the metastatic sites (if present).

Follow up: Patients will continue on androgen deprivation for a total of 2 years. They will be followed clinically and monitored with serum testosterone and Prostate-specific antigen until 2-years after completion of ADT (Androgen deprivation therapy) treatment. Androgen blockade will be the same throughout the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age ≥ 18 years
3. Eastern cooperative oncology group (ECOG) performance status ≤2
4. Documented histologically confirmed adenocarcinoma of the prostate
5. Willing to undergo the following therapy: (1st) Systemic chemo-hormonal therapy with up to 6-months (~24 weeks) of neoadjuvant androgen deprivation and up to 6 cycles of chemotherapy, (2nd) definitive local tumor control with adjuvant radiation therapy, and (3rd) consolidative stereotactic radiation to oligometastatic lesions. Additionally, must be willing to be treated with a full two years of androgen deprivation.
6. Oligometastatic prostate cancer: Stage T1-4, N0-1 and/or M1a-b (up to 5 metastatic lesions- including bone lesions and non-regional lymph nodes seen on bone scan, contrast enhanced CT scan, or positron emission tomography PET scan)

Exclusion Criteria:

1. Prior local non-surgical therapy to treat prostate cancer (e.g. radiation therapy, brachytherapy)
2. Prior therapy to a metastatic site.
3. Prior or ongoing systemic therapy for prostate cancer including, but not limited to:

   1. Hormonal therapy (e.g. leuprolide, goserelin, triptorelin, degarelix)
   2. CYP-17 (cytochrome P450 17α-hydroxy/17,20-lyase) inhibitors (e.g. ketoconazole)
   3. Antiandrogens (e.g. bicalutamide, nilutamide)
   4. Second generation antiandrogens (e.g. enzalutamide, abiraterone)
   5. Immunotherapy (e.g. sipuleucel-T, ipilimumab)
   6. Chemotherapy (e.g. docetaxel, cabazitaxel) *Note: may be enrolled if hormone therapy was recently initiated (<90 days duration)). In the event that hormone therapy was initiated prior to study enrollment, the clock for 2 years of androgen deprivation would begin at the time of therapy initiation, rather than at study enrollment.
4. Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
5. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
6. Abnormal bone marrow function [absolute neutrophil count (ANC)<1500/mm3, platelet count <100,000/mm3, hemoglobin <9 g/dL]
7. Abnormal liver function (bilirubin >ULN ( upper limit of normal); AST (aspartate aminotransferase), ALT (alanine transaminase) > 2.5 x upper limit of normal)
8. Creatinine clearance of ≥ 30 mL/min. CrCl (Creatinine clearance) should be calculated suing the Cockcroft-Gault formula.
9. Active cardiac disease defined as active angina, symptomatic congestive heart failure, or myocardial infarction within previous six months.
10. Prior history of malignancy in the past 3 years with the exception of basal cell and squamous cell carcinoma of the skin. Other malignancies that are considered to have a low potential to progress may be enrolled at discretion of PI.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Pienta, MD, Principal Investigator — SKCCC at Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemohormonal and Definitive Therapy After Prostatectomy
Started | 26
Completed | 25
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemohormonal and Definitive Therapy After Prostatectomy
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 62.2 [55.3 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Assessed by 3-year Prostate-specific Antigen Progression-free Survival Rate
Description: To evaluate efficacy of multimodality therapy in men, defined as the 3 year Prostate-specific antigen progression-free (Prostate-specific antigen<0.2 ng/ml) survival rate among men who have non-castrate testosterone levels 2 years after enrollment.
Time Frame: 3 years
Population: Assessed 25/26 patients (1 patient withdrew from study prior completing TED)
Measure: Count of Participants; unit: Participants
Arm/Group | Chemohormonal and Definitive Therapy After Prostatectomy
Number analyzed (Participants) | 25
Participants
  3-year Prostate-specific antigen PFS (Prostate-specific antigen <0.2), after enrollment | 22
  3-year Prostate-specific antigen PFS (Prostate-specific antigen >=0.2), after enrollment | 3

2. Secondary Outcome: Safety of the 3 Years Multimodality Therapy Assessed Using Common Terminology Criteria for Adverse Events (CTCAE) Version 4 Criteria and the Clavien-Dindo Classification
Description: To assess the safety of multimodality therapy in men presenting with newly diagnosed oligometastatic prostate cancer after prostatectomy. Toxicities related to neoadjuvant therapy, radiation therapy, or stereotactic body radiation therapy (SBRT) will be assessed using CTCAE version 4 criteria. Surgical toxicities will be assessed using the Clavien-Dindo Classification
Time Frame: 3 years
Population: Assessed all patients, from time of enrollment until study exit/3 years from enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemohormonal and Definitive Therapy After Prostatectomy
Number analyzed (Participants) | 26
Participants
  grade 4 neutropenia | 1
  grade 3 neutropenic fever | 1
  No Grades 3 and 4 neutropenia and surgical- or radiation-induced toxicities. | 24

3. Secondary Outcome: Time to Prostate-specific Antigen Recurrence
Description: To investigate the time from an undetectable Prostate-specific antigen (≤0.2 ng/mL) until the Prostate-specific antigen is >0.2 over two time-points.
Time Frame: 3 years
Population: Assessed 25/26 patients (1 patient withdrew from study prior completing TED)
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Chemohormonal and Definitive Therapy After Prostatectomy
Number analyzed (Participants) | 25
Month | NA [NA to NA] — The median time to PSA (Prostate-specific antigen) recurrence within 3 years was not reached because at that timepoint, less than 50% of the participants had experienced a PSA recurrence.

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Chemohormonal and Definitive Therapy After Prostatectomy
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemohormonal and Definitive Therapy After Prostatectomy (N=26)
neutropenia (Blood and lymphatic system disorders) | 1 (1)
neutropenic fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemohormonal and Definitive Therapy After Prostatectomy (N=26)
fatigue (General disorders) | 21 (21)
hot flashes (Vascular disorders) | 10 (10)
neuropathy (Nervous system disorders) | 10 (10)
alopecia; (Skin and subcutaneous tissue disorders) | 5 (5)
dysgeusia (Nervous system disorders) | 5 (5)
hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 4 (4)
skin alterations (Skin and subcutaneous tissue disorders) | 4 (4)
xerosis (Skin and subcutaneous tissue disorders) | 2 (2)
anxiety (Psychiatric disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
edema (lower extremity) (Skin and subcutaneous tissue disorders) | 3 (3)
gastritis (Gastrointestinal disorders) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 3 (3)
gastrointestinal reflux (Gastrointestinal disorders) | 1 (1)
pain (bilateral legs) (Musculoskeletal and connective tissue disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 1 (1)
pain (joint); (Musculoskeletal and connective tissue disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
weight gain (Investigations) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1)
urinary tract obstruction (Renal and urinary disorders) | 1 (1)
oral candidiasis (Gastrointestinal disorders) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
pain (pelvis) (Musculoskeletal and connective tissue disorders) | 1 (1)
memory impairment (Nervous system disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1)
elevated ALT (Investigations) | 1 (1)
elevated AST (Investigations) | 1 (1)
hematochezia (Gastrointestinal disorders) | 1 (1)
xerostomia (Gastrointestinal disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
general body aches (Musculoskeletal and connective tissue disorders) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
epistaxis (Investigations) | 1 (1)
infusion related reaction (Skin and subcutaneous tissue disorders) | 1 (1)
nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
fever (General disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT03043807/Prot_SAP_000.pdf